CLINICAL TRIAL: NCT00428766
Title: A Study of the Safety, Tolerability, and Pharamcokinetics of MORAb-003, a Humanized Monoclonal Antibody, in Subjects With Advanced Ovarian Cancer
Brief Title: Safety, Tolerability and Pharmacokinetics of MORAb-003 in Subjects With Advanced Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Martin Phillips, MD, Morphotek
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-003-001
Record Dates: First submitted 2007-01-28; First posted 2007-01-30 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — farletuzumab

INTERVENTIONS:
Drug: MORAb-003

SUMMARY:
The purpose of this study is to establish the safest dose of MORAb-003 in subjects with advanced ovarian cancer. MORAb-003 is an antibody directed to an antigen on the surface of ovarian cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects, ≥18 years of age, with a histologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal adenocarcinoma, with or without elevation of CA 125, confirmed at the Department of Pathology, Memorial Sloan-Kettering Cancer Center.
2. Subject must have disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) or evaluable by clinical signs/symptoms (e.g., ascites, pleural effusion, or lesions of less than 2 cm) supported by CA-125, radiologic, or pathologic studies conducted within 4 weeks prior to study entry.
3. Subject must have failed at least a standard (platinum-containing) chemotherapy regimen and be considered platinum refractory or resistant.
4. Life expectancy ≥3 months, as estimated by the investigator.
5. Karnofsky performance status ≥70%.
6. Subjects must be surgically sterile, postmenopausal, or using an effective form of contraception.
7. Subjects undergoing treatment with other medications must have been on a stable medication regimen for at least 30 days prior to Study Day 1.
8. Laboratory and clinical results within the 2 weeks prior to Study Day 1 as follows:

   Absolute neutrophil count (ANC) ≥1.5 x 109/L Platelet count ≥100 x 109/L Hemoglobin ≥10 g/dL Serum bilirubin ≤2.0 mg/dL Aspartate transaminase (AST) ≤2.5 x upper limit of normal (ULN) Alanine transaminase (ALT) ≤2.5 x ULN Serum creatinine ≤2.0 mg/dL Amylase ≤1.5 x ULN Lipase ≤1.5 x ULN
9. Spirometry indicating a FEV1 of >79% of predicted.
10. Subject must be willing and able to provide written informed consent.

Exclusion Criteria:

1. Known central nervous system (CNS) tumor involvement.
2. Evidence of other active malignancy.
3. Active asthma or other chronic lung disease.
4. Clinically significant heart disease (e.g., congestive heart failure of New York Heart Association Class III or IV, angina not well controlled by medication, or myocardial infarction within 6 months).
5. ECG demonstrating clinically significant arrhythmias (Note: Subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal SVT, are eligible).
6. Active serious systemic disease, including active bacterial or fungal infection.
7. Chronic inflammatory bowel disease.
8. Chemotherapy, biologic therapy, or immunotherapy within 3 weeks prior to enrollment.
9. Breast-feeding, pregnant, or likely to become pregnant during the study.
10. Active hepatitis or HIV infection.
11. Subjects who have received a previous monoclonal antibody therapy and have evidence of an immune or allergic reaction, or documented HAHA.
12. Subjects with large ascites (≥500 cc based on results of most recent CT scan).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Konner, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States